CLINICAL TRIAL: NCT00710892
Title: CASPALLO: A Phase I Study Evaluating the Use of Allodepleted T Cells Transduced With Inducible Caspase 9 Suicide Gene After Haploidentical Stem Cell Transplantation
Brief Title: CASPALLO: Allodepleted T Cells Transduced With Inducible Caspase 9 Suicide Gene
Acronym: CASPALLO
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21580-CASPALLO
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma; Myelodysplastic Syndrome; Chronic Myeloid Leukemia
Keywords: suicide gene-modified allodepleted donor lymphocytes; given to recipients of haploidentical stem cell transplants; Stage III; Stage IV; Myelodysplastic syndrome; AML after first relapse; primary refractory disease; CML; Hemophagocytic lymphohistiocytosis (HLH); familial hemophagocytic lymphohistiocytosis (FLH); viral-associated hemophagocytic syndrome (VAHS); Severe chronic active Epstein Barr virus infection (SCAEBV); T or NK cell malignancy; X-linked lymphoproliferative disease (XLP)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphohistiocytosis, Hemophagocytic; Histiocytic Sarcoma; Lymphoproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Level 1-3 (Experimental): Administration of suicide gene-modified allodepleted T cells.
  Interventions: Biological: Allodepleted T Cells

INTERVENTIONS:
Biological: Allodepleted T Cells — Dose Level 1 = 1 x 10e6 T cells/kg; Dose Level 2 = 3 x 10e6 T cells/kg; Dose Level 3 = 1 x 10e7 T cells/kg.
  Patients may be enrolled at the next dose level of T cells when all patients at the previous dose level have reached Day 42 post-T cell infusion without unacceptable toxicity.

SUMMARY:
Patients are being asked to participate in this study because they will be receiving a stem cell transplant as treatment for their disease. As part of the stem cell transplant, they will be given very strong doses of chemotherapy, which will kill off all their existing stem cells. Stem cells are created in the bone marrow. They grow into different types of blood cells that we need, including red blood cells, white blood cells, and platelets.

We have identified a close relative of the patients whose stem cells are not a perfect match for the patient, but can be used. This type of transplant is called "allogeneic", meaning that the cells come from a donor. With this type of donor who is not a perfect match, there is typically an increased risk of developing graft-versus-host disease (GvHD) and a longer delay in the recovery of the immune system.

GvHD is a serious and sometimes fatal side effect of stem cell transplant. GvHD occurs when the new donor cells recognize that the body tissues of the patient are different from those of the donor.

In the laboratory, we have seen that cells made to carry a gene called iCasp9 can be killed when they encounter a specific drug called AP1903. To get the iCasp9 into the T cells, we insert it using a virus called a retrovirus that has been made for this study. The drug (AP1903) that will be used to "activate" the iCasp9 is an experimental drug that has been tested in a study in normal donors, with no bad side effects. We hope we can use this drug to kill the T cells. Other drugs that kill or damage T cells have helped GvHD in many studies. However we do not yet know whether AP1903 will kill T cells in humans, even though it has worked in our experimental studies on human cells in animals. Nor do we know whether killing the T cells will help the GvHD. Because of this uncertainty, patients who develop significant GvHD will also receive standard therapy for this complication, in addition to the experimental drug. We hope that having this safety switch in the T cells will let us give higher doses of T cells that will make the immune system recover faster. These specially treated "suicide gene" T cells are an investigational product not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
Because the patient will receive cells with a new gene in them, they will be followed for a total of 15 years to see if there are any long-term side effects of the gene transfer.

Before the conditioning treatment for the transplant, we collected 30 mL (6 teaspoonfuls) of blood from the patient, which we made into a cell line that grows in the laboratory by mixing the blood with a virus called EBV. Some of the cells from this blood were mixed with T cells from the blood stem cell donor, to stimulate cells that might cause GvHD. We then added an investigational agent called RFT5-dgA. The RFT5-dgA helped to get rid of donor T cells that might cause GvHD. To get iCasp9 into the remaining T cells, we have to insert the iCasp9 gene into these cells. This is done with a virus called a retrovirus that has been made for this study, and will carry the iCasp9 gene into the T cells. The virus also has another gene called CD19, which will make the cells express the CD19 protein on their surface. We will not inject the virus directly into the patient, but only into the special T cells we have made in the laboratory. After we have put the virus into the cells, we will select the T cells that have CD19 on their surface, so we know these cells will also have the iCasp9 gene. We will perform tests on the specially treated cells before giving them to the patient, to ensure they only carry the iCasp9 gene, and not the virus itself. This should ensure that no virus can come out of the cells and infect other cells in the body.

TREATMENT PLAN:

To prepare the body for transplantation, the patient will be given high-dose chemotherapy. Further discussion of the treatment plan for the stem cell transplant will be discussed with the patient separately, and they will sign a separate consent form.

If the patient is doing well after the transplant, and they do not have serious GvHD, they will be eligible to receive the special T cells from Day 30 to 90 post-transplant. The specially selected and treated T cells will be given by vein, once. The cells will be given between Day 30 and day 90 after the patient receives their stem cell transplant. We will give special medicines before the IV starts to help prevent allergic reactions that might occur. Because there is a possibility that the specially treated T cells can cause or worsen GvHD, we will not be able to give these cells if the patient already has significant GvHD.

If the patient develops GvHD after being given the specially treated T cells, we will prescribe the new drug that has been shown to kill cells carrying iCasp9. The drug's name is AP1903. It has been tested in normal healthy volunteers, and has not caused any bad effects, but it is not approved by the FDA. Although the drug is not approved by the FDA, the FDA has allowed us to use the drug for this study. This drug will be given as a 2-hour intravenous infusion. We will take 10 mL (2 teaspoonfuls) of blood on days 2, 4, 7 and 14 after the infusion to check if the drug has been successful in killing the specially treated cells. If the patient has mild GvHD, and if the GvHD does not get better with AP1903, we will give the patient additional medicines that are usually used to treat GvHD. If the patient has serious GvHD, we will immediately give additional medicines that are usually used to treat GvHD, as well as AP1903. In some cases though, GvHD does not respond to treatments.

ELIGIBILITY:
INCLUSION CRITERIA:

At the time of transplant:

A. Patients (up to 65 years of age) with:

1. ALL or high grade NHL that is Stage III or IV and has relapsed or is considered to be primary refractory disease.
2. Myelodysplastic syndrome.
3. AML after first relapse or with primary refractory disease.
4. CML
5. Hemophagocytic lymphohistiocytosis (HLH); familial hemophagocytic lymphohistiocytosis (FLH); viral-associated hemophagocytic syndrome (VAHS); patients with severe chronic active Epstein Barr virus infection (SCAEBV) with predilection for T or NK cell malignancy; X-linked lymphoproliferative disease (XLP)

B. Lack of suitable conventional donor (i.e. 5/6 or 6/6 related, or 5/6 or 6/6 unrelated donor) or presence of a rapidly progressive disease not permitting time to identify an unrelated donor.

At the time of allodepleted T cell infusion:

1. Engrafted with ANC greater than 500.
2. Must have greater than or equal to 50% donor chimerism in either peripheral blood or bone marrow, or relapse of their original disease.
3. Life expectancy greater than 30 days
4. Lansky/Karnofsky scores greater than or equal to 60
5. Absence of severe renal disease (creatinine greater than 2X normal for age)
6. Absence of severe hepatic disease (direct bilirubin greater than 2 mg/dL, or SGOT greater than 200
7. Oxygen saturation greater than 94% on room air
8. Patient/Guardian able to give informed consent

EXCLUSION CRITERIA:

At the time of transplant:

1. Pregnancy*

At the time of allodepleted T cell infusion:

1. GvHD
2. Severe intercurrent infection
3. Pregnancy*
4. Other investigational drugs in the prior 30 days

   * Pregnancy test only required for at-risk individuals, defined as female patients of childbearing potential who have received a reduced-intensity conditioning regimen.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum number of suicide gene-modified allodepleted donor lymphocytes that can be given to recipients of haploidentical stem cell transplants that will result in a rate of Grade III/IV GVHD of 25% or less. | 45 days
  Maximum tolerated dose of suicide gene-modified allodepleted donor lymphocytes up to a total of 1 x 10e7/kg per dose.

SECONDARY OUTCOMES:
To evaluate the biological effects of administration of AP1903, a dimerizer used to activate the suicide gene mechanism, and its clinical effects in patients who develop GvHD. | 1 year
  To assess the biological effects (i.e. on numbers of transduced peripheral blood T cells) of AP1903 in patients who develop Grade ≥ I GvHD.
To analyze the contribution of the gene-modified cells to immune reconstitution in these patients by measuring their survival, persistence and expansion. | 15 years
  Investigators will analyze several parameters (Immunophenotyping, T and B cell function) measuring immune reconstitution resulting from iCaspase transduced allodepleted T cells.
To measure the overall and disease-free survival at 100 days and at 1 year post-transplant. | 1 year
  Investigators will measure patients' overall and disease free survival, at 100 days and at 1 year post transplant.
To obtain preliminary information on whether subjects receiving additional doses of cells show a cumulative rise in the percentage of circulating gene-modified cells. | 15 years
  Preliminary information will be obtained on whether patients who receive additional injections of the T cells show a rise in the percentage of circulating gene modified cells.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K Brenner, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang EC, Liu H, West JA, Zhou X, Dakhova O, Wheeler DA, Heslop HE, Brenner MK, Dotti G. Clonal Dynamics In Vivo of Virus Integration Sites of T Cells Expressing a Safety Switch. Mol Ther. 2016 Apr;24(4):736-45. doi: 10.1038/mt.2015.217. Epub 2015 Dec 7. PMID 26639404
- [Derived] Zhou X, Di Stasi A, Brenner MK. iCaspase 9 Suicide Gene System. Methods Mol Biol. 2015;1317:87-105. doi: 10.1007/978-1-4939-2727-2_6. PMID 26072403
- [Derived] Zhou X, Di Stasi A, Tey SK, Krance RA, Martinez C, Leung KS, Durett AG, Wu MF, Liu H, Leen AM, Savoldo B, Lin YF, Grilley BJ, Gee AP, Spencer DM, Rooney CM, Heslop HE, Brenner MK, Dotti G. Long-term outcome after haploidentical stem cell transplant and infusion of T cells expressing the inducible caspase 9 safety transgene. Blood. 2014 Jun 19;123(25):3895-905. doi: 10.1182/blood-2014-01-551671. Epub 2014 Apr 21. PMID 24753538
- [Derived] Di Stasi A, Tey SK, Dotti G, Fujita Y, Kennedy-Nasser A, Martinez C, Straathof K, Liu E, Durett AG, Grilley B, Liu H, Cruz CR, Savoldo B, Gee AP, Schindler J, Krance RA, Heslop HE, Spencer DM, Rooney CM, Brenner MK. Inducible apoptosis as a safety switch for adoptive cell therapy. N Engl J Med. 2011 Nov 3;365(18):1673-83. doi: 10.1056/NEJMoa1106152. PMID 22047558